CLINICAL TRIAL: NCT02791776
Title: Impact of the Choice of the Distal Vertebral When Posterior Instrumentation in the Surgery of the Thoracic Adolescent Idiopathic Scoliosis
Brief Title: Impact of the Choice of the Distal Vertebral in the Surgery of the Thoracic Adolescent Idiopathic Scoliosis
Acronym: VD-SIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-HPNCL-04
Record Dates: First submitted 2016-06-01; First posted 2016-06-07 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-06

CONDITIONS: Scoliosis
Keywords: scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Scoliosis (Other): self-administered questionnaire (SRS 30) to assess the state of health and disability of patients.
  collection of patient's radiographic and clinical parameters
  Interventions: Other: Scoliosis

INTERVENTIONS:
Other: Scoliosis — self-administered questionnaire (SRS 30) to assess the state of health and disability of patients.
  Collection of patient's radiographic and clinical parameters

SUMMARY:
The problem of choosing the supporting vertebra was the subject of several studies. They do not suggest as regards the techniques that are not currently used or with insufficient setback.

The need to have a sufficient number of files with a minimum decline of 5 years for proposing a multicenter study that will be conducted within the framework of the Scoliosis Research Group (SRG) and will result in a roundtable at the next congress GES in March 2015. the GES gathers most of the teams that support this pathology.

DETAILED DESCRIPTION:
Idiopathic scoliosis is a deformity in three planes of space the child's spine and scalable teenager with growth. In adults is causing severe deformities of respiratory failure responsible and disabling back pain. Scoliosis is most often idiopathic without cause found that the genetic origin is being identified. It is detected by the school doctor, the doctor or pediatrician. The management is based primarily on monitoring small angle discoveries scoliosis and the orthopedic treatment of progressive scoliosis by the specialized services of pediatric orthopedics or rehabilitation as recommended by the HAS (February 2008). Surgical treatment is reserved for the orthopedic treatment failures or advanced scoliosis discovered too late.

The goal of surgery is to reduce as much as possible distortion in the three planes of space and avoid the progression of the deformity in adulthood. Its principle is to correct the deformity using instrumentation and maintain over time this correction with a bone graft. This is commonly called spinal fusion with instrumentation. The instrumentation includes all of the vertebral anchors connected to rods.

Indications are asked in each case most often in adolescence and sometimes in younger children and rarely in adulthood. The procedure performed in adolescence allows to benefit from a flexible spine still allowing good reduction of the deformation, a lesser neurological risk and good consolidation of the bony fusion guarantees a stable income in the long term.

Among all types of curves, thoracic scoliosis pose the problem of choosing the bends to be instrumented. This choice is an essential element for the initial correction and become the long-term. It is the result of a compromise between a long instrumentation that orchestrates all of the deformation to the detriment of the mobility of the lumbar spine and a shorter instrumentation that preserves mobility at the expense perhaps of a smaller reduction. These short instrumentations called selective thoracic instrumentation, the choice of the support or lower vertebra vertebra of instrumentation is an unsolved problem and is the subject of this work.

The immediate results of the posterior vertebral arthrodesis are assessed by the correction of the deformity in three planes of space: measuring the angle of the curvature in the coronal plane, analyzing the return of a physiological kyphosis in sagittal plane and correction of the vertebral rotation in the horizontal plane. The results for medium and long term are assessed by analyzing the maintenance of correction of the deformity and the evolution of the above spine and above underlying arthrodesis. This is appreciated by the coronal and sagittal balance, changing the supporting vertebra and the first non-instrumented vertebra and evolution spine underlying uninstrumented.

The problem of choosing the supporting vertebra was the subject of several studies. They do not suggest as regards the techniques that are not currently used or with insufficient setback.

The need to have a sufficient number of files with a minimum decline of 5 years for proposing a multicenter study that will be conducted within the framework of the Scoliosis Research Group (SRG) and will result in a roundtable at the next congress GES in March 2015. the GES gathers most of the teams that support this pathology.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic idiopathic scoliosis (Lenke 1 or 2) of the child in puberty and adolescent surgery for posterior spinal fusion with instrumentation with a minimum decline of 5 years.
* Thoracic scoliosis Lenke 1 or 2.
* Affiliates or beneficiaries of a social security scheme
* Initial medical examination.

Exclusion Criteria:

* Scoliosis adult scoliosis and whose age at the time of the transaction is less than 10 years.
* Double major scoliosis (Lenke 3 or 4)
* Scoliosis thoracolumbar or lumbar (Lenke 5 or 6).
* Non-idiopathic scoliosis.
* Opposition by the patient or legal guardian with the use of pre- and postoperative data

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 157 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Analyze at least up of 5 years, the development of the first non-instrumented vertebra and spine underlying depending on the choice of the supporting vertebra thoracic idiopathic scoliosis adolescents who underwent selective thoracic instrumentation. | Comparaison beetween before the chirurgical intervention and 5 years later
  The results should be assessed using the position of the distal vertebra of the instrumentation with respect to the neutral vertebra. The distal vertebra will be identified VN if it matches the neutral vertebra, VN-1, VN-2 ... if it is located above the VN and VN + 1, TN + 2 ... to a vertebra situated below the vertebra neutral.

SECONDARY OUTCOMES:
Evaluate the impact of this correction on the quality of life of patients with self-administered questionnaire (SAQ Parent, patient SAQ) | Comparaison beetween before the chirurgical intervention and 5 years later
  SRS 30 questionnaires scores.
To evaluate the incidence and predictors of complications. | Comparaison beetween before the chirurgical intervention and 5 years later
  Incidence and predictors of complications factors
To evaluate the influence of the correction of the deformity | Comparaison beetween before the chirurgical intervention and 5 years later
  % Reduction in primary and secondary curvatures

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc CLEMENT, MD, Principal Investigator — Fondation LENVAL, Hôpitaux Pédiatriques de Nice CHU-LENVAL
Locations (16):
- France (15):
  - Institut François Calot/Centre Hélio-Marin, Berck
  - Groupe hospitalier Pellegrin, Bordeaux
  - HFME, Lyon
  - Hôpital de la Timone Enfants, Marseille
  - CHU Hôpital Nord, Marseille
  - Chirurgie infantile, Hôpital mère-enfant pédiatrie, CHU Nantes, Nantes
  - Fondation LENVAL, Hôpitaux Pédiatriques de Nice CHU-LENVAL, Nice
  - Hôpital Saint-Joseph, Paris
  - APHP - Hôpital Necker-Enfants-Malades, Paris
  - AP-HP Hôpital Robert Debré, Paris
  - Clinique Chirurgicale Infantile, Hôpital Charles Nicolle, CHU de Rouen, Rouen
  - Groupe Hospitalier Sud Réunion Terre Rouge Boissy, Saint-Pierre
  - CHU Hôpital des Enfants, Toulouse
  - CHU de Tours Hôpital Clocheville, Tours
  - Centre du rachis, Maison de Spécialistes de Trélazé, sur le site du Village Santé Angers Loire, Trélazé
- Hotel Dieu De France Hospital Youssef Souda, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No